CLINICAL TRIAL: NCT04706975
Title: A Randomized, Double-blind, Placebo-controlled, Proof-of-concept Study to Evaluate the Efficacy and Safety of Oral Difelikefalin (CR845) for Moderate to Severe Pruritus in Adult Subjects With Notalgia Paresthetica
Brief Title: Study to Evaluate the Efficacy and Safety of Oral Difelikefalin (CR845) for Moderate to Severe Pruritus in Subjects With Notalgia Paresthetica (KOMFORT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845-210601
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Pruritus; Notalgia Paresthetica
Keywords: Notalgia Paresthetica; Pruritus; CR845; Chronic Itch; difelikefalin; Itch; Itching; Generalized pruritus; NP; Neuropathic itch
MeSH Terms: conditions — Pruritus | interventions — difelikefalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Difelikefalin 2.0 mg (Active Comparator): Oral difelikefalin 2.0 mg tablet administered twice daily
  Interventions: Drug: difelikefalin 2.0 mg
- Placebo (Placebo Comparator): Oral placebo tablet administered twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: difelikefalin 2.0 mg — Oral difelikefalin 2.0 mg administered twice daily
  Other Names: CR845
  Arms: Difelikefalin 2.0 mg
Drug: Placebo — Oral Placebo administered twice daily
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of twice-daily (BID) oral difelikefalin (CR845) in adult subjects with notalgia paresthetica and moderate to severe pruritus.

DETAILED DESCRIPTION:
The study will consist of a 37-day Screening period, a 7-day Run-In period, a 8-week Placebo-Controlled Treatment period followed by a 4-week Active Extension period and a Follow Up visit approximately 14 days after the last dose of study drug.

All subjects will sign an informed consent form (ICF) and undergo screening for study eligibility.

Subjects will be randomized to receive either placebo or difelikefalin (CR845) tablets at a dose of 2.0 mg, orally BID. Intake of the first dose of study drug will be at Day 1.

Subjects who complete the Placebo-Controlled Treatment period of the study will transition into the Active Extension period upon completion of the Week 8 visit assessments. All subjects in the Active Extension will receive difelikefalin (CR845).

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible for inclusion into the study, a patient must meet the following criteria:

* Subject has clinically confirmed diagnosis of active Notalgia Paresthetica;
* Subject has a history of chronic pruritus due to Notalgia Paresthetica;
* Subject has moderate to severe pruritus;
* Female subject is not pregnant or nursing during any period of the study.

Key Exclusion Criteria:

A patient will be excluded from the study if any of the following criteria are met:

* Subject has pruritus attributed to a cause other than Notalgia Paresthetica;
* Subject has any clinically significant medical condition or physical/laboratory/ECG/vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the weekly mean of the daily 24-hour Worst Itch-Numeric Rating Scale (WI-NRS) score at Week 8. | Baseline, Week 8

SECONDARY OUTCOMES:
Improvement in itch-related quality of life as assessed by the change from baseline to Week 8 in total Skindex-10 Scale score | Baseline, Week 8
Change from baseline in itch-related Sleep Disturbance Subscale measured by the Itch Medical Outcomes Study (MOS) at Week 8 | Baseline, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Nilam Shah, Study Director — Cara Therapeutics
Locations (36):
- United States (26):
  - Cara Therapeutics Study Site, Fort Smith, Arkansas
  - Cara Therapeutics Study Site, Hot Springs, Arkansas
  - Cara Therapeutics Study Site, Rogers, Arkansas
  - Cara Therapeutics Study Site, Fountain Valley, California
  - Cara Therapeutics Study Site, Los Angeles, California
  - Cara Therapeutics Study Site, San Diego, California
  - Cara Therapeutics Study Site, Santa Monica, California
  - Cara Therapeutics Study Site, Cromwell, Connecticut
  - Cara Therapeutics Study Site, Coral Gables, Florida
  - Cara Therapeutics Study Site, Margate, Florida
  - Cara Therapeutics Study Site, Miami, Florida
  - Cara Therapeutics Study Site, North Miami Beach, Florida
  - Cara Therapeutics Study Site, Sandy Springs, Georgia
  - Cara Therapeutics Study Site, Indianapolis, Indiana
  - Cara Therapeutics Study Site, Plainfield, Indiana
  - Cara Therapeutics Study Site, Metairie, Louisiana
  - Cara Therapeutics Study Site, New York, New York
  - Cara Therapeutics Study Site, High Point, North Carolina
  - Cara Therapeutics Study Site, Columbus, Ohio
  - Cara Therapeutics Study Site, Charleston, South Carolina
  - Cara Therapeutics Study Site, Bellaire, Texas
  - Cara Therapeutics Study Site, Pflugerville, Texas
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site, Salt Lake City, Utah
  - Cara Therapeutics Study Site, Norfolk, Virginia
  - Cara Therapeutics Study Site, Spokane, Washington
- Canada (10):
  - Cara Therapeutics Study Site, Surrey, British Columbia
  - Cara Therapeutics Study Site, Winnipeg, Manitoba
  - Cara Therapeutics Study Site, Markham, Ontario
  - Cara Therapeutics Study Site, Peterborough, Ontario
  - Cara Therapeutics Study Site, Montreal, Quebec
  - Cara Therapeutics Study Site, Markham
  - Cara Therapeutics Study Site, Montreal
  - Cara Therapeutics Study Site, Peterborough
  - Cara Therapeutics Study Site, Surrey
  - Cara Therapeutics Study Site, Winnipeg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim BS, Bissonnette R, Nograles K, Munera C, Shah N, Jebara A, Cirulli J, Goncalves J, Lebwohl M; KOMFORT Trial Investigators. Phase 2 Trial of Difelikefalin in Notalgia Paresthetica. N Engl J Med. 2023 Feb 9;388(6):511-517. doi: 10.1056/NEJMoa2210699. PMID 36780675